CLINICAL TRIAL: NCT01366391
Title: Therapeutic Monitoring of Metformin in Women With Polycystic Ovary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biocinese (Industry)
Responsible Party: Naura Tonin Angonese, Biocinese
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0038.0 208.00-09
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-06

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; metformin; pharmacokinetic
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Other): study parallel with one arm only.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin 500 mg tablet (1000 or 1500 mg/day)
  Other Names: Glifage 500 mg

SUMMARY:
Metformin is one of the most commonly prescribed drugs worldwide for the treatment of Type 2 Diabetes. It has been currently used for the treatment of: polycystic ovary syndrome, gestational diabetes, metabolic syndrome and obesity. In patients with polycystic ovary syndrome (PCOS) the adverse side effects are a frequent cause for treatment discontinuation. In every day medical practice lower doses of Metformin are administered searching for the continuation of the treatment.

However, there is no clinical study to support this assertion. The objective of this study is to monitor and correlate the therapeutic effect of Metformin on patients with PCOS taking daily doses of 1500mg and 1000mg.

DETAILED DESCRIPTION:
Patients with PCOS diagnosis and that are able to attempt the inclusion criteria are divided in two groups: administration of metformin 500 mg tablet three times/day as well 1500 mg/day (group A)and administration of metformin 500 mg tablet twice/day or 1000 mg/day (group B). Blood samples were collected to the pharmacokinetic evaluation from first day of administration until 3 months after beginning of treatment. The patients are monitored during 3 months and all side effects are register. The efficacy of both treatment are analyzed by biochemical and physical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 40 years old, with no use of contraceptive drugs or insulin sensitizing agents for more than 3 months.
* PCOS diagnosis.
* Insulin resistance Index by the Homeostatic model Assessment Formula higher than 2.5.

Exclusion Criteria:

* Another diseases with androgen excess;
* Patients with history of serious adverse reaction or hypersensibility to any medicine;
* History or presence of renal, hepatic or gastrointestinal disorders.
* Continuous use of any pharmaco, inclusively metformin

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-08 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of metformin | First day after administration until 3 months after begining of treatment
  Blood samples are collected from each patient and the plasma concentration is analysed.

SECONDARY OUTCOMES:
Number of adverse events | observation during 3 months of treatment
  All adverse events are registered during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Naura Angonese, Dr, Principal Investigator — Biocinese
Locations (1):
- Biocinese, Toledo, Paraná, Brazil